CLINICAL TRIAL: NCT07262515
Title: Integrative Epidemiology of Prognosis in Patients With Acute Alcoholic Hepatitis at AP-HP
Acronym: DIONYSOS
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: DAT23012
Record Dates: First submitted 2025-11-17; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-09

CONDITIONS: Acute Alcoholic Hepatitis
Keywords: Acute Alcoholic Hepatitis; Machine Learning; Accelerated failure time; RWE epidemiology; Prognosis prediction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute alcoholic hepatitis: All adult patients diagnosed with acute alcoholic hepatitis at AP-HP hospitals, identified using ICD-10 codes (K701), pathology reports, and clinical data.

SUMMARY:
Acute alcoholic hepatitis (AAH) is a severe liver disease that often occurs in individuals with prolonged excessive alcohol consumption. Patients face a high risk of liver failure, complications, and death, despite available treatments. Current prognostic scores based on blood tests provide limited accuracy and do not capture the full complexity of the disease.

The purpose of this study is to improve the prediction of patient outcomes after a diagnosis of acute alcoholic hepatitis. By integrating clinical, biological, and histological information collected from the AP-HP data warehouse, the investigators aim to identify more reliable prognostic markers. This could help physicians better tailor treatments and improve survival of patients affected by this condition.

DETAILED DESCRIPTION:
Acute alcoholic hepatitis (AAH) is characterized by acute liver inflammation caused by prolonged excessive alcohol intake. It is associated with jaundice, liver failure, and in severe cases, multi-organ failure and death. Current prognostic scores rely primarily on serum biomarkers of liver function but fail to account for systemic complications or histological features.

This retrospective, multicenter observational study conducted at AP-HP hospitals will analyze a large cohort of patients diagnosed with AAH since 2017. Data extracted from the AP-HP Clinical Data Warehouse (EDS) will include demographics, comorbidities, biological markers (liver and renal function tests, coagulation parameters, lactate), histological findings (necrosis, fibrosis, neutrophil infiltration, bilirubinostasis), microbiology results, prescribed medications, and outcomes such as infections, need for liver transplantation, and mortality.

The primary outcome is overall survival after diagnosis. Secondary outcomes include the impact of intermediate factors such as bacterial or fungal infections, alcohol withdrawal, organ failure, and transplantation on prognosis. Statistical analyses will combine classical survival models (Cox regression, Accelerated Failure Time models) and modern machine learning approaches (random forest, gradient boosting).

The goal is to develop integrative prognostic models that provide a more accurate and personalized assessment of prognosis in AAH, ultimately guiding clinical decision-making and improving patient management.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years)
* Diagnosis of acute alcoholic hepatitis (ICD10 K701 or occurrence of the terms "HAA" (French translation of "AAH" or "hépatite alcoolique aiguë" (French translation of "acute alcoholic hepatitis") in a pathology report, followed by manual verification

Exclusion Criteria:

- Patients younger than 18 years at diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with acute alcoholic hepatitis across all AP-HP hospitals. Data will be collected retrospectively from the AP-HP Clinical Data Warehouse (EDS).
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival after diagnosis of acute alcoholic hepatitis | From diagnosis up to 7 years after
  Overall survival will be assessed using mortality data recorded in the AP-HP Clinical Data Warehouse. The objective is to evaluate prognosis and identify risk factors associated with death after a diagnosis of acute alcoholic hepatitis, by integrating clinical, biological, and histological information. Survival will be analysed at multiple time points, including 1 month, 6 months, and 1 year after diagnosis.

SECONDARY OUTCOMES:
Incidence of bacterial or fungal infections after diagnosis | Within 7 years after diagnosis
  Evaluate the impact of bacterial or fungal infections occurring after diagnosis of acute alcoholic hepatitis on the risk of death
Requirement for liver transplantation | Within 7 years after diagnosis
  Evaluate the influence of the need for liver transplantation after diagnosis of acute alcoholic hepatitis on the risk of death
Organ failure occurrence | within 7 years after diagnosis
  Evaluate the impact of organ failure following a diagnosis of acute alcoholic hepatitis on the risk of death
Impact of alcohol withdrawal on prognosis | within 7 years after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Vincent MALLET, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Necker Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No